CLINICAL TRIAL: NCT03106766
Title: A Single-center, Double-blind, Controlled Study to Evaluate the Effect of Next Science™ Acne Cream on Mild to Moderate Facial Acne in Adult Females Over 6 Months.
Brief Title: Six Months Evaluation of Next Science Acne Creams on Facial Acne in Adult Females.
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Decision from the Sponsor
Sponsor: Next Science TM (Industry)
Collaborators: Skin Laser & Surgery Specialists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSP-004
Record Dates: First submitted 2017-03-27; First posted 2017-04-10 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acne cream 1x (Experimental): Twice-daily facial applications of the 1X product (avoiding contact with eyes and all mucous membranes) to the entire face for 6 months.
  Interventions: Drug: Acne cream 1X
- Acne cream 2x (Experimental): Twice-daily facial applications of the 2X product (avoiding contact with eyes and all mucous membranes) to the entire face for 6 months.
  Interventions: Drug: Acne cream 2X

INTERVENTIONS:
Drug: Acne cream 2X — Twice daily application of facial acne cream 2X after facial cleansing
  Arms: Acne cream 2x
Drug: Acne cream 1X — Twice daily application of facial acne cream 1X after facial cleansing
  Arms: Acne cream 1x

SUMMARY:
To assess facial acne vulgaris clinical and psychological outcomes by measuring differences in lesions counts, investigator global assessment, and subjects quality of life scores over 6 months in adult females treated with Next Science™ acne cream 2x or Next Science™ acne cream 1x in a double blind manner.

DETAILED DESCRIPTION:
This is a 6-month, single-site, double-blind, controlled study in 20 female subjects with mild to moderate facial acne. Subjects will be randomized 1:1 to apply either topical Next Science™ acne cream 2x or Next Science™ acne cream 1x daily. Subjects will be evaluated for clinical acne and quality of life outcomes at baseline, 6, 12, 18 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female ages 18 and above
2. Has 20 or more inflammatory lesions on the face (papules and pustules) as determined by qualified examiner at Start of Treatment.
3. In the area to be treated, has no significant facial dermatological conditions other than acne (as determined by the investigator) that would interfere with any study treatment or procedure
4. Is willing and able to discontinue use of all baseline acne treatments for the duration of their trial participation
5. Agrees to refrain from professional facial treatments during their trial participation.
6. Agrees to avoid tanning booth use and minimize sun exposure during their trial participation.
7. Is willing and able to follow instructions and procedures including attending scheduled study visits, which will require adequate transportation to the study site
8. Is able to read, understand and sign the informed consent document and communicate with study staff and investigator.

Exclusion Criteria:

1. Has more than 2 nodules/cystic acne lesions on the face
2. Has a history of significant reactions to topical acne treatments, or a known allergy or hypersensitivity to any listed ingredients
3. Has any history of skin malignancy
4. Has used any systemic medications (including antibiotics, estrogens, retinoids) primarily for treatment of acne in the 21 days prior to randomization.
5. Has used estrogens primarily as treatment for acne in the 21 days prior to randomization (estrogens prescribed for other reasons will be allowed if stable for at least 30 days prior to randomization).
6. Has had any professional facial treatments in the 14 days prior to randomization.
7. Has received any investigational treatment in the 30 days prior to randomization.
8. Have any significant medical problems or other issues that would, in the investigator's judgment, affect their suitability for participation in this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Reduction in Lesion Count | Baseline versus 6 months
  Inflammatory acne lesions with both study acne cream products after 6 months of treatment compared to baseline. This will be measured as the mean percent change from baseline to week 24 in the inflammatory lesion count.

SECONDARY OUTCOMES:
Inflammatory Lesion count over time | weeks 6, 12, 18, and 24
  to assess the mean percent change from baseline to weeks 6, 12, 18, and 24 inflammatory lesion counts
Non-inflammatory acne lesion over time | weeks 6, 12, 18, and 24
  to assess the mean percent change from baseline to weeks 6, 12, 18, and 24 in non-inflammatory lesion counts
Investigator Global Assessment over time | weeks 6, 12, 18, and 24
  to assess the mean percent change from baseline to weeks 6, 12, 18, and 24 in IGA
Treatment Areas over time | weeks 6, 12, 18, and 24
  to assess the mean percent change from baseline to weeks 6, 12, 18, and 24 in treatment areas (erythema, dryness, stinging or burning, erosion, edema, pain and itching)
Quality of Life over time | weeks 6, 12, 18, and 24
  The Acne-QoL questionnaire containing 19 questions organized into four domains which address the impact of facial acne on health-related quality of life will be administered. These are Self Perception, Role-social, Role-emotional and Acne Symptoms. Results will assess the mean percent change from baseline to weeks 6, 12, 18, and 24 in QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Myntti, PhD, Study Director — Next Science
Locations (1):
- Skin Laser & Surgery Specialists of NY & NJ, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marshall-Hudson A, Tuley M, Damstra M, Dosik JS, Myntti MF, Porral D, Palomo J. A 6-month, Multi-center, Double-blind, Controlled Study to Evaluate the Effect of a Biofilm Disrupting Acne Cream on Mild-to-Moderate Facial Acne in Female Volunteer Subjects. J Clin Aesthet Dermatol. 2023 Apr;16(4):43-52. PMID 37077927